CLINICAL TRIAL: NCT02087813
Title: A Single Center Open Label Pilot Study of Alpha1-Antitrypsin: A Novel Treatment to Mitigate Neuromyelitis Optica Attacks
Brief Title: Pilot Study of alpha1-antitrypsin to Treat Neuromyelitis Optica Relapses
Acronym: A1AT for NMO
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-27176
Record Dates: First submitted 2014-03-11; First posted 2014-03-14 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Neuromyelitis Optica
Keywords: neuromyelitis optica; optic neuritis; longitudinally extensive transverse myelitis
MeSH Terms: conditions — Neuromyelitis Optica; Optic Neuritis | interventions — alpha 1-Antitrypsin; Methylprednisolone; Methylprednisolone Hemisuccinate

ARMS (2):
- A1AT (Experimental): Alpha1-antitrypsin 120mg/kg once weekly for a total of 4 doses, to be given intravenously. This will be given in addition to standard of care 3-5 days of 1000mg IV methylprednisolone.
  Interventions: Drug: Alpha1-antitrypsin; Drug: methylprednisolone
- Standard of care (Active Comparator): Patients that do not wish to receive study treatment but agree to otherwise follow study protocol will also be enrolled in an observational cohort. They will receive the standard of care 3-5 days 1000mg IV methylprednisolone.
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: Alpha1-antitrypsin
  Other Names: ARALAST NP; alpha1-proteinase inhibitor
  Arms: A1AT
Drug: methylprednisolone — 3-5 days 1000mg IV methylprednisolone at first presentation with acute attack.
  Other Names: Solu-Medrol

SUMMARY:
Neuromyelitis Optica (NMO) is a rare, devastating demyelinating disease of the central nervous system (CNS) that has different causes and treatments from the more common demyelinating disease multiple sclerosis (MS). Current NMO therapies are nonspecific and have varying and often suboptimal benefit. The investigators will evaluate whether use of alpha1-antitrypsin (A1AT, an FDA-approved medication for patients with congenital deficiency of A1AT associated with emphysema) can benefit acute attacks of NMO, improving patient disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Age ≥18 and ≤ 75 years.
* Diagnosis of NMO or NMO spectrum disorder (NMOSD). The diagnosis of NMO will conform to the 2006 Wingerchuk criteria.1, 2 The diagnosis of NMOSD will include patients with relapsing optic neuritis and aquaporin-4 antibody (AQP4) seropositivity or patients with relapsing longitudinally extensive transverse myelitis and AQP4 seropositivity.2-5 NMO and NMOSD will be collectively referred to as NMO.
* AQP4-antibody positivity.
* Present with an acute NMO attack (see definition below).
* Patients must not have a history of clinically significant infusion reactions with administration of biologic agents.
* If on chronic treatment for NMO, treatment was initiated at least 3 months earlier and medication dose is stable. Additional restrictions will be placed on changes in concomitant symptomatic medications.
* A female subject of childbearing potential must have a negative serum pregnancy test at the screening visit and agree to use a medically reliable method of contraception (e.g., barrier with either spermicide or hormonal contraception) until study completion.
* Agree to answer the questions on the Columbia Suicide Severity Rating Scale at each specified visit.

Exclusion Criteria:

* A woman who is pregnant, breastfeeding, or planning pregnancy.
* If the patient is enrolled in any other experimental trial or on other experimental therapy.
* If the patient has a known IgA deficiency with IgA-antibodies.
* Any medical condition or clinically significant laboratory abnormality that in the Investigator's judgment may affect the patient's ability to safely complete the study.

Acute attack:

* The occurrence of new or worsening neurological symptoms consistent with optic neuritis, transverse myelitis, or a brain lesion that develop acutely (i.e., patients must present within 7 days of symptom onset).
* The symptoms must persist for at least 48 hours, are not attributable to confounding clinical factors (e.g., fever, infection, injury, adverse reactions to concomitant medications).
* The symptoms must be accompanied by sensory, motor or visual acuity objective deficits, which must be verified by the examining physician.
* A single episode of a paroxysmal symptom (e.g., tonic spasm) is not a relapse; however, the new onset of multiple occurrences of a paroxysmal symptom over at least 48 hours can be a relapse if accompanied by a new, corresponding objective deficit.
* Sensory symptoms with no change on clinical examination, fatigue, mood change, or bladder or bowel urgency or incontinence will not be sufficient to establish a relapse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in disability from baseline/nadir to week 24 as assessed by Opticospinal Impairment Score (OSIS) subscale. | Baseline, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.

SECONDARY OUTCOMES:
Mean change in disability from baseline/nadir to week 24 as assessed by Expanded Disability Status Scale (EDSS). | Baseline, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.
For patients experiencing optic neuritis, mean change in visual acuity from baseline/nadir to week 24 as assessed by Sloan 2.5% low contrast visual acuity chart. | Baseline, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.
Mean change in retinal nerve fiber layer from baseline/nadir to week 24 as assessed by optical coherence tomography (OCT). | Baseline and Week 24
Mean change in length of spinal cord lesion from baseline/nadir to week 24 as assessed by magnetic resonance imaging (MRI) T2 sequences. | Baseline, Week 24

OTHER OUTCOMES:
Suicidality as a Measure of Safety and Tolerability | Screening, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.
  Columbia Classification Algorithm for Suicide Assessment (C-SSRS).
Serum biomarkers, including cytokines, elastase level, A1AT level, neutrophil elastase activity. | Baseline, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.
Cerebral Spinal Fluid (CSF) biomarkers, including neurofilament, GFAP, MBP, neutrophil elastase activity, A1AT level, cytokines. | Baseline and Week 8
  Lumbar puncture.
Quality of life as a Measure of Safety and Tolerability | Baseline, Week 1: Day 2, Week 2, 3, 4, 8, 16, and 24.
  Functional Assessment of Multiple Sclerosis Quality of Life instrument (FAMS).
Electrocardiogram (ECG) as a Measure of Safety and Tolerability | Baseline, Day 2, and Week 16.
Urinalysis as a Measure of Safety and Tolerability | Baseline, Day 2, and Week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Goodyear, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States